CLINICAL TRIAL: NCT05099458
Title: Characterization of Molecular Signature Associated With T-cell Dysfunction Observed During Chronic HBV Infection
Brief Title: T-cell Dysfunction in Chronic HBV Infection
Acronym: VHB-Roche
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6847
Record Dates: First submitted 2018-11-23; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Hepatitis B Virus
Keywords: T lymphocytes; Exhaustion; Molecular signature
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatitis B (Experimental)
  Interventions: Biological: Additional blood sampling (100 ml)

INTERVENTIONS:
Biological: Additional blood sampling (100 ml) — only an additional blood volume will be collected at the same time of the standard blood collection for these patients

SUMMARY:
Chronic hepatitis B (CHB) infection remains an important public health with more than 240 million people chronically infected despite the existence of an effective vaccine. Cirrhosis and hepatocellular carcinoma (HCC) are major complications of CHB infection and are responsible for more than 600,000 deaths each year. These complications are strongly related to the function of the immune system. Indeed, the persistence of HBV and the progression of liver disease are mainly due to the development of an ineffective immune response to HBV. Therefore, the clinical outcome depends on the complex interaction between HBV replication and adaptive immune responses.

The ultimate goal of antiviral treatments is the elimination of HBsAgHBs and the appearance of anti-HBs antibodies without detectable PCR replication. Current treatments are effective at lowering viral DNA levels, but they are not able to permanently eliminate chronic HBV infection, due to the persistence of cDNA in the nucleus of infected hepatocytes. This therapeutic goal is rarely achieved and new therapeutic approaches are needed. In this sense, Immunotherapy represents a very promising new therapeutic approach that could lead to the cure of chronic HBV infection. Indeed, HBV infection is characterized by a progressive depletion of T lymphocytes which results in a progressive loss of function, associated with a sustained positive regulation of inhibitory control molecules.

Thus, the objective of this study is to define the immune signature and the main control pathways associated with T-cell depletion in patients chronically infected with HBV, by analyzing immune cells isolated from these patients at phenotypic , transcriptional and functional levels

ELIGIBILITY:
Inclusion Criteria:

1. For all patients

   * Compensated liver disease defined by the following criteria: Conjugated bilirubin level ≤ 1.2 x upper limit of normal (ULN), TP / INR ≤ 1.2 × ULN, platelets ≥ 150 x 109 / L, serum albumin ≥ 35 g / L, and no history of clinical hepatic decompensation (ascites, jaundice, encephalopathy, variceal hemorrhage) (results from a blood test dating up to 8 months before inclusion).
   * Adequate haematological function: platelets ≥ 150x109 / L, Hb ≥ 12 g / dL (male) or ≥ 11 g / dL (female), white blood cells ≥4x109 / L and <11x109 / L, except for ethnic neutropenia (these values must be obtained at least 8 months before inclusion)
   * Male or female between 20 and 69 years of age, inclusive
   * 18.5 ≤BMI ≤ 35 kg / m²
   * Patients who dated and signed informed consent
2. For patients chronically infected with NUC treatment for more than 6 months:

   * HBV DNA <25 IU / mL
   * HBsAg-positive (≥100 IU / mL)
   * HBeAg-negative or positive
   * ALT <1.5x ULN
3. For chronically infected, untreated patients:

   * HBsAg positive (≥100 IU / mL)
   * negative or positive HBeAg
   * HBV DNA> 2000 IU / mL
   * ALT <2 x ULN

Exclusion Criteria:

* Use of steroids or other immunosuppressive agents that would affect the number and / or function of immune cells in the last 4 weeks

  •,Any disease or other major medical disorder or condition that , that, in the judgment of the investigator, would interfere with results of the study (including, but not limited to: cancer, systemic lupus erythematosus, rheumatoid arthritis or other autoimmune disease, etc. ...)
* Major surgery or traumatic injury (including blood transfusion) in the last 4 weeks

  -• Use of an experimental drug in the last 12 weeks
* Positive test for Hepatitis C, HIV, Hepatitis D, or Hepatitis A (anti-HAV IgM) at the time of inclusion
* Significant acute infection such as influenza or other clinically significant illness in the last 2 weeks
* History of drug abuse in the last year
* positive pregnancy test for women of childbearing age
* Breast-feeding women
* Patients presenting:

  1. a medical history or signs of cirrhosis defined by a biopsy result or any other non-invasive validated test showing cirrhosis, OR
  2. Either during the selection visit: a transient elastography value ≥ 10.5 kPa OR a Fibrotest® / Fibrosure® score ≥ 0.48 and an APRI score ≥1 .

Note: If a biopsy or a non-invasive test for cirrhosis has never been performed in the patient, then the medical examinations described in b) must be performed during the selection visit.

* History of ascites, digestive hemorrhage and / or encephalopathy
* Any co-morbidity that could lead to liver damage as judged by the investigator (excessive alcohol consumption, hemochromatosis, Wilson's disease, autoimmune hepatitis, inflammatory colitis ...)
* Patients unable or unwilling to comply with the protocol requirements
* Patient unable to give informed consent

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-04-25 (Estimated); Study Completion 2022-04-25 (Estimated)

PRIMARY OUTCOMES:
Phenotypic analyze of exhausted T-cells (CD4 and CD8) | Day 0
  a blood sample will be analysed to see the impact of chronic HBV infection on T cell dysfunction.
Transcriptional analyze of exhausted T-cells (CD4 and CD8) | Day 0
  a blood sample will be analysed to see the impact of chronic HBV infection on T cell dysfunction.

SECONDARY OUTCOMES:
Response to functional T-cells stimulation tests | Day 0
  This response will be evaluated by functional T cell stimulation tests in the presence or absence of immunomodulatory molecules targeting immune checkpoint receptors such as PD1, but also Tim-3, LAG3 or others.

CONTACTS AND LOCATIONS:
Overall Officials: François HABERSETZER, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Hopitaux Universitaires de Strasbourg, Strasbourg, France